CLINICAL TRIAL: NCT02999477
Title: A Pilot Study Of Changes In PD-L1 Expression During Preoperative Treatment With Nab-Paclitaxel And Pembrolizumab In Hormone Receptor-Positive Breast Cancer
Brief Title: A Study Of Changes In PD-L1 Expression During Preoperative Treatment With Nab-Paclitaxel And Pembrolizumab In Hormone Receptor-Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adrienne G. Waks (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Adrienne G. Waks, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-466
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Results first posted 2024-09-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nab-Paclitaxel (Experimental): * 2 weeks Nab-Paclitaxel Run in
  * Biopsy will be performed
  * Post mono therapy Nab-Paclitaxel administered weekly
  * Post mono therapy Pembrolizumab administered every 3 weeks
  * Agents administered for a total of 15 weeks
  Interventions: Drug: Pembrolizumab; Drug: Nab-Paclitaxel; Procedure: Biopsy
- Pembrolizumab (Experimental): * 2 weeks Pembrolizumab Run in
  * Biopsy will be performed
  * Post mono therapy Nab-Paclitaxel administered weekly
  * Post mono therapy Pembrolizumab administered every 3 weeks
  * Agents administered for a total of 14 weeks
  Interventions: Drug: Pembrolizumab; Drug: Nab-Paclitaxel; Procedure: Biopsy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered in clinic every three weeks.
  Other Names: Keytruda
Drug: Nab-Paclitaxel — Nab-Paclitaxel will be administered in clinic every week.
  Other Names: Abraxane
Procedure: Biopsy — Biopsies for research purposes will be performed at three separate timepoints during treatment.

SUMMARY:
This research study is exploring chemotherapy in combination with immunotherapy (a therapy that uses the body's own immune system to control cancer) as a possible treatment for hormone receptor positive breast cancer.

The interventions involved in this study are:

* Pembrolizumab (MK-3475; Keytruda™)
* Nab-Paclitaxel (Abraxane

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study intervention.

In this research study, the investigators are looking at how the participants body and tumor respond to the combination of Nab-paclitaxel and Pembrolizumab. Also, the investigators will be examining the participants tumor tissue to learn more about the disease.

The FDA (the U.S. Food and Drug Administration) has not approved Pembrolizumab for this specific disease; but it has been approved in the United States for the treatment of other diseases.

The FDA has not approved Nab-paclitaxel as a treatment option for this type of breast cancer; but it has been approved in the United States for the treatment of metastatic breast cancer (breast cancer that has spread to other parts of the body).

Pembrolizumab is a medicine that may treat cancer by working with the participant's immune system. The immune system is the body's natural defense against disease. The immune system sends types of cells called "T cells" throughout the body to detect and fight infections and diseases, including cancer. For some types of cancer, the T cells do not work as they should and are prevented from attacking the tumors. Pembrolizumab is thought to work by blocking a protein in the T cells called PD-1 ("programmed death 1"), which then allows these cells and other parts of the immune system to attack tumors.

Nab-paclitaxel (Abraxane) is part of a class of medications called antimicrotubule agents. It works by stopping the growth and spread of cancer cells by blocking the action of proteins called microtubules.

The combination of Pembrolizumab and Nab-paclitaxel is investigational. "Investigational" means that the combination of study drugs is being studied. The study drugs, when given separately, work in different ways to stop the cancer cells from growing and spreading. However, it is not known if giving the two study drugs at the same time will have a better anti-cancer effect than giving each treatment on its own.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive breast cancer.
* Participants must have operable breast cancer, with tumors greater than or equal to 2 cm in size; Participants must not have any evidence of distant metastatic disease. Inflammatory breast cancer is permitted.
* All confirmed invasive disease must have been tested for ER, PR, and HER2 and participants must have hormone receptor-positive, HER2-negative breast cancer (ER>1% or PR>1%, AND HER2-negative per ASCO CAP guidelines, 2013).
* Participants with multicentric, multifocal, and/or contralateral cancers are allowed as long as one lesion meets eligibility and no biopsied tumor is HER2+.
* Prior systemic therapy: No prior chemotherapy, biologic therapy, hormonal therapy or investigational therapy for this operable breast cancer.
* Prior radiation therapy: No prior radiation to the ipsilateral breast.
* The participant is ≥18 years old
* The participant has an Eastern Cooperative Oncology Group (ECOG) performance status ≤1 (see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1500/mm3
  * Platelets ≥100,000/mm3
  * Hemoglobin ≥9 g/dL
  * Total Bilirubin ≤1.5 mg/dL (< 2.0 in participants with known Gilbert's syndrome)
  * Serum creatinine ≤1.5 mg/dL OR calculated GFR ≥60mL/min
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal.
  * International normalized ratio (INR) or Prothrombin Time (PT) <1.5 times the upper limit of normal unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
  * Activated Partial Thromboplastin Time (aPTT) <1.5 times the upper limit of normal unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* The participant is capable of understanding and complying with the protocol and has signed the informed consent document.
* The participant must be willing to undergo the three required research biopsies over the course of protocol therapy. Participants who undergo an attempted research biopsy procedure for the purpose of this protocol, and in whom inadequate tissue is obtained, are not required to undergo a repeat biopsy in order to continue on protocol.
* The effects of pembrolizumab on the developing human fetus are unknown. For this reason, both women and men of child-bearing potential must agree to use adequate contraception (Section 5.5.2) starting with the first dose of study therapy and for the duration of study participation, through 120 days after the last dose of study medication.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. While on the study, women may not breast-feed. Women of childbearing potential are defined as those who have not been surgically sterilized or have not been free from menses for > 1 year.

* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Participants on bisphosphonates may continue receiving bisphosphonate therapy during study treatment.

Exclusion Criteria:

* The participant has received prior pembrolizumab or any other anti-PD-1, anti-PD-L1, or anti-PD-L2 therapy, or has participated in any prior studies involving pembrolizumab
* Hypersensitivity to pembrolizumab or any of its excipients.
* The participant has any history or evidence of active, non-infectious pneumonitis or interstitial lung disease.
* The participant has an uncontrolled intercurrent illness including, but not limited to, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, congestive heart failure (New York Heart Association Class III or IV; see Appendix B), active ischemic heart disease, myocardial infarction within the previous six months, uncontrolled diabetes mellitus, chronic liver or renal disease, or severe malnutrition.
* Concurrent use of potent CYP3A4 inhibitors (see Appendix C), such as ketoconazole and erythromycin, should be avoided during the study treatment with nab-paclitaxel.
* Pregnant women are excluded from this study because pembrolizumab has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab, breastfeeding should be discontinued if the mother is treated with pembrolizumab.
* Active infection requiring intravenous antibiotics at week 1 day 1.
* Individuals with a history of a second malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and non-melanoma cancer of the skin. Participants with other cancers diagnosed within the past 5 years and felt to be at low risk of recurrence should be discussed with the study sponsor to determine eligibility.
* The participant has a medical condition that requires chronic systemic steroid therapy or any other form of immunosuppressive medication including disease modifying agents, or has required such therapy in the last 2 years. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* The participant has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents.
* The participant is known to be positive for Hepatitis B surface antigen, or Hepatitis C RNA. Testing for screening is not required.
* Known HIV-positive participants.HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pembrolizumab. In addition, these participants are at increased risk of lethal infections with bone marrow suppressive therapy, i.e. nab-paclitaxel. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated. Testing for screening is not required.
* The participant has received a live vaccine within 28 days of planned start of study therapy.
* Seasonal influenza vaccines for infection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (i.e. Flu-Mist ®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2026-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Gropper Waks, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fu J, Waks AG, Pimenta E, Titchen B, Bi K, Camp S, Pappa T, Keenan T, Shannon E, Vigneau S, Bemus M, Nag A, Thorner AR, Park J, DiLullo M, Wrabel E, Jeselsohn R, Mittendorf EA, Abravanel DL, Tolaney SM, Van Allen EM. Cellular reprogramming during anti-PD-1 and chemotherapy treatment in early-stage primary hormone receptor-positive breast cancer. Nat Commun. 2025 Nov 28;16(1):10704. doi: 10.1038/s41467-025-66659-y. PMID 41315371
- [Result] Waks AG, Fu J, Chu X, Binboga Kurt B, Li T, Kuntz TM, Shen Y, Yang D, Meli K, Reardon B, Park J, Partridge A, Abravanel D, Jeselsohn R, Wrabel E, Alberti J, DiLullo M, Chen S, Mohammed-Abreu A, Sun X, Balko JM, Kleijn M, Audeh W, Morgan XC, Krop IE, Tayob N, Van Allen EM, Mittendorf EA, Tolaney SM. Efficacy, safety, and predictive biomarkers of neoadjuvant nab-paclitaxel and pembrolizumab in hormone receptor-positive breast cancer: A randomized pilot trial. Nat Commun. 2025 Nov 28;16(1):10705. doi: 10.1038/s41467-025-66667-y. PMID 41315271

RESULTS

PARTICIPANT FLOW:
Groups:
- Nab-Paclitaxel: * 2 weeks Nab-Paclitaxel Run in
  * Biopsy will be performed
  * Post mono therapy Nab-Paclitaxel administered weekly
  * Post mono therapy Pembrolizumab administered every 3 weeks
  * Agents administered for a total of 15 weeks
  Pembrolizumab: Pembrolizumab will be administered in clinic every three weeks.
  Nab-Paclitaxel: Nab-Paclitaxel will be administered in clinic every week.
  Biopsy: Biopsies for research purposes will be performed at three separate timepoints during treatment.
- Pembrolizumab: * 2 weeks Pembrolizumab Run in
  * Biopsy will be performed
  * Post mono therapy Nab-Paclitaxel administered weekly
  * Post mono therapy Pembrolizumab administered every 3 weeks
  * Agents administered for a total of 14 weeks
  Pembrolizumab: Pembrolizumab will be administered in clinic every three weeks.
  Nab-Paclitaxel: Nab-Paclitaxel will be administered in clinic every week.
  Biopsy: Biopsies for research purposes will be performed at three separate timepoints during treatment.
Period: Overall Study
Arm/Group | Nab-Paclitaxel | Pembrolizumab
Started | 16 | 16
Completed | 15 | 14
Not Completed | 1 | 2
Not completed — found ineligible after first dose | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nab-Paclitaxel | Pembrolizumab | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Median (Full Range); unit: years] | 46 [31 to 70] | 41.5 [31 to 53] | 42 [31 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 14 | 12 | 26
  Race: Asian | 0 | 2 | 2
  Race: More than one race | 1 | 0 | 1
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Non-Hispanic | 13 | 13 | 26
  Unknown | 1 | 1 | 2
ECOG PS = 0 at Baseline [Count of Participants; unit: Participants] — The ECOG PS scale indicates increasing levels of disability, with 0 indicating fully active; 1, restricted in strenuous activity; 2, restricted in work activity but ambulatory and capable of self-care; 3, capable of limited self-care; 4, completely disabled; and 5, dead
  Participants | 15 | 14 | 29
Stage [Count of Participants; unit: Participants] — Stage refers to the extent of your cancer, such as how large the tumor is and if it has spread.The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Participants
    II | 10 | 10 | 20
    III | 5 | 4 | 9
T Stage [Count of Participants; unit: Participants] — T followed by a number from 0 to 4 describes the main (primary) tumor's size and if it has spread to the skin or to the chest wall under the breast. Higher T numbers mean a larger tumor and/or wider spread to tissues near the breast.
  Participants
    T2 | 10 | 10 | 20
    T3 | 4 | 4 | 8
    T4 | 1 | 0 | 1
N Stage [Count of Participants; unit: Participants] — NX: The lymph nodes were not evaluated.
  N0: Either:
  No cancer was found in the lymph nodes. Only areas of cancer smaller than 0.2 mm are in the lymph nodes. N1: The cancer has spread to 1 to 3 axillary lymph nodes and/or the internal mammary lymph nodes. If the cancer in the lymph node is larger than 0.2 mm but 2 mm or smaller, it is called "micrometastatic" (N1mi).
  N2: The cancer has spread to 4 to 9 axillary lymph nodes. Or, it has spread to the internal mammary lymph nodes, but not the axillary lymph nodes.
  Participants
    N0 | 5 | 3 | 8
    N1 | 10 | 11 | 21
Hormone receptor status [Count of Participants; unit: Participants]
  ER+/PR- | 3 | 1 | 4
  ER+/PR+ | 9 | 8 | 17
  ER+/PR low+ | 1 | 2 | 3
  ER low+/PR- | 2 | 3 | 5
HER2 status [Count of Participants; unit: Participants]
  negative | 15 | 14 | 29
  positive | 0 | 0 | 0
Size of breast tumor by physical exam (cm) [Median (Full Range); unit: cm] | 4 [2 to 7] | 5 [2 to 15] | 4.5 [2 to 15]
Histology [Count of Participants; unit: Participants]
  Ductal | 11 | 11 | 22
  Lobular | 3 | 1 | 4
  Both | 1 | 2 | 3
Grade [Count of Participants; unit: Participants] — Grade is usually described using a number from 1 to 3 or 4. The higher the number, the more different the cancer cells look from healthy cells and the faster they are growing.
  Participants
    1 | 1 | 1 | 2
    2 | 7 | 7 | 14
    3 | 7 | 5 | 12
    Unknown | 0 | 1 | 1
Contralateral invasive breast ca at diagnosis [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 14 | 14 | 28
Breast surgery [Count of Participants; unit: Participants]
  Lumpectomy | 6 | 6 | 12
  Mastectomy | 8 | 8 | 16
  No breast surgery | 1 | 0 | 1
Adjuvant radiation [Count of Participants; unit: Participants]
  Yes | 11 | 7 | 18
  No | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in the Biomarker (PD-L1) Expression
Description: PDL1 H-Score by Immunohistochemistry (≥ 100 versus 0-99) change from baseline biopsy to biopsy after 2-week monotherapy (from C1D1 to C3D1).
  The minimum score is 0 and the higher the score the worse.
Time Frame: 2 weeks
Population: Patients with biomarker sample available at both C1D1 and C3D1 time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel | Pembrolizumab
Number analyzed (Participants) | 11 | 12
Participants
  <100 | 11 | 12
  >=100 | 0 | 0
Statistical Analysis 1: Comparison: Nab-Paclitaxel; Test type: Equivalence — The null hypothesis is no change in the amount of PD-L1 expression from baseline to after a two-week run in of nabpaclitaxel. The test was using one-sided alpha (type I error) of 0.05. The margin is zero; p = 1.0, McNemar
Statistical Analysis 2: Comparison: Pembrolizumab; Test type: Equivalence — The null hypothesis is no change in the amount of PD-L1 expression from baseline to after a two-week run in of nabpaclitaxel or pembrolizumab. The test was using one-sided alpha (type I error) of 0.05; p = 1.0, McNemar

2. Secondary Outcome: Change in Percentage of Stromal Tumor Infiltrating Lymphocytes After Monotherapy Treatment
Description: stromal tumor infiltrating lymphocytes (sTIL) is measured at C1D1 and C3D1 of the treatment.
Time Frame: from C1D1 to C3D1 (2 weeks)
Population: We are including patients who have biopsy both at C1D1 and C3D1.
Measure: Mean (Full Range); unit: percentage of stromal TILs
Arm/Group | Nab-Paclitaxel | Pembrolizumab
Number analyzed (Participants) | 10 | 10
percentage of stromal TILs | 7.2 [-65 to 60] | 0.5 [-10 to 15]

3. Secondary Outcome: Pathologic Complete Response Rate
Description: Response is measured by RCB score.RCB 0 (equal to pCR), RCB I(minimal burden), RCB II (moderate burden) and RCB III(extensive burden)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel | Pembrolizumab
Number analyzed (Participants) | 15 | 14
Participants | 2 | 1

4. Secondary Outcome: Overall Response Rate
Description: Overall response rate, assessed radiographically by both Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) following treatment with combination nab-paclitaxel and pembrolizumab in the neoadjuvant setting. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the baseline LD. Overall response = CR+PR+SD
Time Frame: 2 years
Population: 19 patients (9 in Arm A and 10 in Arm B) who had MRI scans during study.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel | Pembrolizumab
Number analyzed (Participants) | 9 | 10
Participants | 7 | 8

5. Secondary Outcome: Disease-Free Survival
Description: Disease-free survival (DFS) will be defined from the time of randomization until the occurrence of the first of the following events:
  * Local/regional recurrence: a recurrent or new invasive ipsilateral breast cancer, invasive breast cancer in the axilla, regional lymph nodes, chest wall, or skin of the ipsilateral breast.
  * Contralateral invasive breast cancer,
  * Distant recurrence: metastatic disease that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer. A single new lesion on a bone scan without evidence of lytic disease on x-ray and without symptoms does not in and of itself constitute distant recurrence, but multiple new bone lesions, or increased isotope uptake associated with new bone symptoms are more likely due to metastases. Bone metastases must be documented with x-rays and clinical description.
  * Death from any cause
Time Frame: 3 years from randomization
Measure: Number (95% Confidence Interval); unit: percentage of DFS patients
Arm/Group | Nab-Paclitaxel | Pembrolizumab
Number analyzed (Participants) | 15 | 14
percentage of DFS patients | 92 [79 to 100] | 100 [100 to 100]

ADVERSE EVENTS:
Time Frame: From randomization as early as 2017-06-02 to post surgery evaluation as late as 2022-10-27. (5 years and 4 months)
Description: The analysis population for mono therapy (nab) excluded two untreated patients. The analysis population for mono therapy (pem) excluded two untreated patients. The analysis population for combination (nab+pem) excluded three untreated patients.
Groups:
- Nab-Paclitaxel Run in: * 2 weeks Nab-Paclitaxel Run in
  * Biopsy will be performed
  Pembrolizumab: Pembrolizumab will be administered in clinic every three weeks.
  Nab-Paclitaxel: Nab-Paclitaxel will be administered in clinic every week.
  Biopsy: Biopsies for research purposes will be performed at three separate timepoints during treatment.
- Pembrolizumab Run in: * 2 weeks Pembrolizumab Run in
  * Biopsy will be performed
  Pembrolizumab: Pembrolizumab will be administered in clinic every three weeks.
  Nab-Paclitaxel: Nab-Paclitaxel will be administered in clinic every week.
  Biopsy: Biopsies for research purposes will be performed at three separate timepoints during treatment.
- Post Monotherapy Nab-Paclitaxel and Pembrolizumab: * Post mono therapy Nab-Paclitaxel administered weekly
  * Post mono therapy Pembrolizumab administered every 3 weeks
  Pembrolizumab: Pembrolizumab will be administered in clinic every three weeks.
  Nab-Paclitaxel: Nab-Paclitaxel will be administered in clinic every week.
Arm/Group | Nab-Paclitaxel Run in | Pembrolizumab Run in | Post Monotherapy Nab-Paclitaxel and Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 1/29
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 4/29
Other Adverse Events (participants affected / at risk) | 6/15 | 1/15 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel Run in (N=15) | Pembrolizumab Run in (N=15) | Post Monotherapy Nab-Paclitaxel and Pembrolizumab (N=29)
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel Run in (N=15) | Pembrolizumab Run in (N=15) | Post Monotherapy Nab-Paclitaxel and Pembrolizumab (N=29)
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 8
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 5
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Fever (General disorders) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 4
Blurred vision (Eye disorders) | 0 | 0 | 2
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hot flashes (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT02999477/Prot_SAP_001.pdf